CLINICAL TRIAL: NCT04358731
Title: A Phase 2/3, Randomized, Observer-blind, Controlled, Multi-Center Study to Evaluate the Lot to Lot Consistency of SIIPL Meningococcal ACYWX Conjugate Vaccine (NmCV-5) and to Compare Its Safety and Immunogenicity With That of Licensed Meningococcal ACWY Vaccine Menactra® in Healthy Individuals 18-85 Years of Age
Brief Title: Study to Evaluate the Lot to Lot Consistency of SIIPL Meningococcal ACYWX Conjugate Vaccine and to Compare Its Safety and Immunogenicity With That of Licensed Meningococcal ACWY Vaccine Menactra® in Healthy Individuals 18-85 Years of Age
Acronym: ACYWX-04
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Serum Institute of India Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ACYWX-04
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-03

CONDITIONS: Vaccine for Meningococcal Disease
MeSH Terms: interventions — NmCV-5 vaccine; Meningococcal Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NmCV-5 (Experimental): A total of 1640 subjects 18 to 85 years of age will be accrued contemporaneously across three age groups - 18 to 29 years, 30 to 60 years, and 61 to 85 years.
  Within each age group subjects will be randomly assigned in a 3:1 ratio to receive either NmCV-5 or Menactra.
  The NmCV-5 subjects in 18-29 year age group will be further randomized 1:1:1 into three different lots (Lot A, B & C) of NmCV-5.
  Total 1230 subjects will be enrolled in NmCV-5 arm.
  Interventions: Biological: NmCV-5
- Menactra (Active Comparator): Subjects will be randomly assigned in a 3:1 ratio to receive either NmCV-5 or Menactra.
  In Menactra arm, total 410 subjects will be enrolled.
  Interventions: Biological: Menactra

INTERVENTIONS:
Biological: NmCV-5 — The NmCV-5 is a fixed-combination available as the lyophilized powder containing meningococcal groups A and X polysaccharides conjugated to tetanus toxoid and meningococcal groups C, W and Y polysaccharides conjugated to CRM197 protein. The vaccine will be reconstituted with normal saline just prior to administration.
  The NmCV-5 lyophilized powder component contains sucrose, sodium citrate and trometamol as excipients. This component is presented as a freeze-dried powder in a single dose vial. No preservative or adjuvant is present in the vaccine.
  The normal saline diluent is a sterile clear colorless liquid in a single dose glass ampoule.
  Arms: NmCV-5
Biological: Menactra — The control vaccine is the licensed meningococcal serogroups ACYW conjugate vaccine (Menactra), manufactured by Sanofi Pasteur Incorporated. Menactra is supplied as a single 0.5 mL dose formulated in sodium phosphate buffered isotonic sodium chloride solution to contain 4 mcg each of meningococcal A, C, Y, and W polysaccharides conjugated to approximately 48 mcg of diphtheria toxoid protein carrier. No preservative or adjuvant is added during manufacture.
  Arms: Menactra

SUMMARY:
This is a Phase 2/3, randomized, observer blind, multi-centre, controlled study to evaluate the safety, immune response and consistency of immune response of three consecutively manufactured lots of NmCV-5 in healthy individuals between the ages of 18 to 85 years (both inclusive). The immune response of NmCV-5 will also be statistically compared against a licensed conjugate vaccine against ACYW (Menactra).

A total of 1640 subjects 18 to 85 years of age will be accrued contemporaneously across three age groups - 18 to 29 years, 30 to 60 years, and 61 to 85 years. Within each age group subjects will be randomly assigned in a 3:1 ratio to receive either NmCV-5 or Menactra. The NmCV-5 subjects in 18-29 year age group will be further randomized 1:1:1 into three different lots (Lot A, B & C) of NmCV-5.

All the randomized subjects will receive a single dose of 0.5 ml of NmCV-5 or Menactra on Day 1. Post vaccination site visits are planned on Days 8, 29 and 180 and a telephonic call at Day 85.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female 18 through 85 years of age, both inclusive, at the time of study vaccine administration.
2. Provide written informed consent.
3. The subject is resident of the study area and is willing to comply with study protocol requirements, including availability for all scheduled visits of the study.
4. Healthy, as determined by medical history and clinical assessment of the investigator.
5. Female subjects of childbearing potential must have a negative urine pregnancy test within 24 hours prior to study vaccine administration.

Exclusion Criteria:

1. Acute illness, at the time of study vaccine administration (once acute illness is resolved, if appropriate, as per investigator assessment, subject will be re-revaluated for eligibility).
2. History of any meningococcal vaccine administration.
3. Current or previous, confirmed or suspected disease caused by N. meningitidis.
4. Household contact with and/or intimate exposure to an individual with any laboratory confirmed N. meningitidis infection within 90 days prior to vaccination.
5. History of severe allergic reactions after previous vaccinations or hypersensitivity to any study vaccine component including tetanus, diphtheria and diphtheria toxoid (CRM197).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1640 (Actual)
Dates: Start 2019-12-27 (Actual); Primary Completion 2021-03-24 (Actual); Study Completion 2021-03-24 (Actual)

PRIMARY OUTCOMES:
rSBA assay Geometric Mean Titers (GMTs) at Day 29 against serogroups A, C, W, Y and X in subjects 18 to 29 years of age. | 1 month after vaccination
Percentage of subjects with seroresponse 28 days after vaccination in pooled NmCV-5 and Menactra vaccine groups | 28 days after immunization

SECONDARY OUTCOMES:
rSBA GMTs at Days 1 and 29 against serogroups A, C, W, Y and X in pooled NmCV-5# and Menactra vaccine groups. | Days 1 and 29

CONTACTS AND LOCATIONS:
Overall Officials: Dr Prasad Kulkarni, MD, Study Director — Serum Institute of India Pvt. Ltd.
Locations (11):
- India (11):
  - Kempegowda Institute of Medical Sciences (KIMS) Hospital & Research Centre, K. R. Road, V. V. Puram, Bangalore 560004, Karnataka, India, Bangalore, Karnataka
  - M S Ramaiah Medical College and Hospitals, Bangalore, Bangalore, Karnataka
  - T. N. Medical College and B. Y. L. Nair Charitable, Mumbai, Maharashtra
  - Seth G S Medical College & KEM Hospital, Mumbai, Maharashtra
  - Jahangir Clinical Development Centre Pvt. Ltd., Pune, Pune, Maharashtra
  - KEM Hospital Research Centre, Vadu Rural Health Program, Vadu Budruk, Taluka - Shirur, District - Pune 412216 , Maharashtra Pune, Pune, Maharashtra
  - Department of community Medicine, Dr Sushila Nayar School of Public Health, Mahatma Gandhi Institute of Medical Sciences, Sewagram, Wardha, Maharashtra
  - Hamdard Institute of Medical Sciences and Research (HIMSR), and Associated Hakeen Abdul Hameed Centenary Hospital (HAHCH) Jamia Hamdard, Hamdard Nagar, New Delhi - 110062, New Delhi, National Capital Territory of Delhi
  - Institute of Medical Sciences and SUM Hospital Bhubaneshwar, Bhubaneshwar, Odisha
  - Sri Ramachandra Institute of Higher Education and Research, Chennai, Tamil Nadu
  - Post Graduate Institute of Medical Education and Research (PGIMER), Chandigarh

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: After one year of study completion

REFERENCES:
- [Derived] Kulkarni PS, Kawade A, Kohli S, Munshi R, Maliye C, Gogtay NJ, S RH, Singh K, Vengadakrishnan K, Panigrahi SK, Sahoo J, Bavdekar A, Garg BS, Raut A, Raj JP, Saxena U, Chaudhari VL, Patil R, Venkatarao E, Kumari N, Surendran J, Parulekar V, Gagnon L, Gensale T, Dharmadhikari A, Gairola S, Kale S, Pisal SS, Dhere RM, Mallya A, Poonawalla CS, Kapse D. Safety and immunogenicity of a pentavalent meningococcal conjugate vaccine versus a quadrivalent meningococcal conjugate vaccine in adults in India: an observer-blind, randomised, active-controlled, phase 2/3 study. Lancet Infect Dis. 2025 Apr;25(4):399-410. doi: 10.1016/S1473-3099(24)00576-0. Epub 2024 Nov 6. PMID 39521012